CLINICAL TRIAL: NCT01121003
Title: Effects of a Weight Maintenance, High Fructose Diet and of Exercise on Hepatic Lipid Metabolism
Brief Title: Effects of Fructose and Exercise on Hepatic Lipid Metabolism
Acronym: FRUCTEXER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor of Physiology, University of Lausanne
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Protocole 220/09
Record Dates: First submitted 2010-05-06; First posted 2010-05-11 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Metabolism
Keywords: Fructose; VLDL-triglycerides; de novo lipogenesis; Human metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low fructose diet/no exercise (Other)
  Interventions: Behavioral: weight maintenance, low sugar diet
- high fructose diet/no exercise (Experimental)
  Interventions: Behavioral: weight maintenance, high fructose diet
- high fructose diet+exercise (Experimental)
  Interventions: Behavioral: weight maintenance, high fructose diet+ exercise

INTERVENTIONS:
Behavioral: weight maintenance, low sugar diet
  Arms: Low fructose diet/no exercise
Behavioral: weight maintenance, high fructose diet
  Arms: high fructose diet/no exercise
Behavioral: weight maintenance, high fructose diet+ exercise
  Arms: high fructose diet+exercise

SUMMARY:
8 healthy male volunteers will be studied each on 3 occasions, ie

* after 4 days on a weight maintenance diet containing 5% simple sugars + low physical activity
* after 4 days on a weight maintenance diet containing 30% fructose + low physical activity
* after 4 days on a weight maintenance diet containing 30% fructose + high physical activity At the end of each of these 3 periods, fructose induced hepatic de novo lipogenesis (13C palmitate synthesis in response to ingestion of a 13C fructose load) and plasma VLDL-triglyceride kinetics (measured with a bolus of 2H-labeled glycerol) will be measured

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 30 years
* males
* BMI between 19 and 25
* low to moderate physical activity (< 3 sessions/week)

Exclusion Criteria:

* smoking
* consumption of alcohol>50g/week
* consumption of drugs or illicit substances
* food allergies

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Hepatic de novo lipogenesis | after 4 days on controlled diet+exercise
  Measurement of 13C VLDL palmitate after ingestion of 13C fructose

SECONDARY OUTCOMES:
Plasma VLDL-triglyceride kinetics | after 4 days on controlled diet+exercise
  Modelling of 2H5-glycerol incorporation in VLDL afetr administration of a bolus of 2H5 glycerol

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — University of Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland